CLINICAL TRIAL: NCT00202748
Title: Phase 3 Study of Changing of Lifestyle by Persons in Risk of Type 2 Diabetes
Brief Title: Change of Lifestyle by Persons in Risk of Type 2 Diabetes
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sorlandet Hospital HF (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SSHF70201
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2005-12-23 (Estimated); Status verified 2003-12

CONDITIONS: Type 2 Diabetes
Keywords: metabolic syndrome; lifestyle; obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Metabolic Syndrome; Obesity

INTERVENTIONS:
Behavioral: Increase in activity to control weight
Behavioral: Increase in activity to control weight.

SUMMARY:
We know that changing lifestyle can prevent type 2 diabetes. The challenge is how to help people changing their lifestyle. We have people in 2 groups: half of them is meeting in grops of 10 persons (interventiongroup), the other ones are just visiting their doctor (controlgroup).

DETAILED DESCRIPTION:
The intervention group are meeting different healt proffesionals (nurse, doctor, eksperts on nutrition,experts on activity and experts on how to change. They have 7 meetings in groups of 10 persons over 3 months. The controlgroup are just meeting their own doctor or the doctor in the hospital 2 times a year.

We tell all that small changes are making big differenses (in weight and the chanse of getting ill). Everyone is told that lack of aktivity is the main reason to obesity. Lack of activity also influense in whar you eat. herefore is activity in the "center".

ELIGIBILITY:
Inclusion Criteria: Diabetes risk score above 9 points.

Exclusion Criteria: Persons with diabetes, serious heart disease, cancer or psychiatric disorder. They have to speak and understand Norwegian language.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220
Dates: Start 2004-03; Study Completion 2007-03

PRIMARY OUTCOMES:
Weigtreduction
Increase in maximum oxygen uptake
Change in foodintake
Change in self-reported activity

SECONDARY OUTCOMES:
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Frode Gallefoss, Dr., Study Chair
Locations (1):
- Sorlandet Hospital, Kristiansand, Serviceboks 416, Norway

REFERENCES:
- [Derived] Nilsen V, Bakke PS, Rohde G, Gallefoss F. Is sense of coherence a predictor of lifestyle changes in subjects at risk for type 2 diabetes? Public Health. 2015 Feb;129(2):155-61. doi: 10.1016/j.puhe.2014.12.014. Epub 2015 Feb 13. PMID 25682903
- [Derived] Nilsen V, Bakke PS, Rohde G, Gallefoss F. Predictors of health-related quality of life changes after lifestyle intervention in persons at risk of type 2 diabetes mellitus. Qual Life Res. 2014 Nov;23(9):2585-93. doi: 10.1007/s11136-014-0702-z. Epub 2014 May 1. PMID 24789668
- [Derived] Nilsen V, Bakke PS, Gallefoss F. Effects of lifestyle intervention in persons at risk for type 2 diabetes mellitus - results from a randomised, controlled trial. BMC Public Health. 2011 Nov 25;11:893. doi: 10.1186/1471-2458-11-893. PMID 22117618